CLINICAL TRIAL: NCT00980343
Title: A Biomarker and Phase II Study of GDC-0449 in Patients With Recurrent Glioblastoma Multiforme
Brief Title: GDC-0449 in Treating Patients With Recurrent Glioblastoma Multiforme That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02922; NCI-2012-02922 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000654829; ABTC-0904 (Other: Adult Brain Tumor Consortium); ABTC-0904 (Other: CTEP); U01CA137443 (NIH)
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (pre-surgery vismodegib) (Experimental): Patients receive oral Hedgehog antagonist GDC-0449 (vismodegib) once daily for 7 days before therapeutic conventional surgery. Beginning within 28 days after surgical resection, all patients receive oral Hedgehog antagonist GDC-0449 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study; laboratory biomarker analysis
  Interventions: Drug: vismodegib; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (no vismodegib pre-surgery) (Experimental): Patients do not receive treatment before therapeutic conventional surgery.
  Beginning within 28 days after surgical resection, all patients receive oral Hedgehog antagonist GDC-0449 (vismodegib) once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other: laboratory biomarker analysis
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vismodegib — Given orally
  Other Names: Erivedge; GDC-0449; Hedgehog antagonist GDC-0449
  Arms: Arm I (pre-surgery vismodegib)
Procedure: therapeutic conventional surgery — undergo surgery
Other: laboratory biomarker analysis — correlative studies
Other: pharmacological study — correlative studies
  Arms: Arm I (pre-surgery vismodegib)

SUMMARY:
This randomized phase II trial is studying how well GDC-0449 works in treating patients with recurrent glioblastoma multiforme that can be removed by surgery. GDC-0449 may be effective in treating patients with glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. 6-month progression-free survival (PFS-6) measured from start of treatment following surgery.

SECONDARY OBJECTIVES:

I. Toxicity. (Clinical) II. Overall survival. (Clinical) III. Tumor response. Partial Response (PR) + Complete Response (CR): MacDonald criteria). (Clinical)

Correlative Studies

* Determination of in vivo drug effect in recurrent Glioblastoma Multiform (GBM). (Correlative studies)
* Determination of in vitro drug effect on CD133+ glioma-derived neurospheres. (Correlative studies)
* Determination of Sonic Hedgehog pathway activation in primary vs. recurrent GBM. (Correlative studies)

TERTIARY OBJECTIVES:

I. Correlate clinical outcome (6 mo PFS) with biologic correlates (1-3) above.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral Hedgehog antagonist GDC-0449 once daily for 7 days before surgery.

Arm II: Patients do not receive treatment before surgery. Beginning within 28 days after surgical resection, all patients receive oral Hedgehog antagonist GDC-0449 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Fresh and paraffin-embedded tissue samples are collected for correlative laboratory studies.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven glioblastoma which is progressive or recurrent following radiation therapy +/- chemotherapy
* Patients must have measurable contrast-enhancing progressive or recurrent glioblastoma by MRI imaging prior to starting treatment; patient must be able to tolerate MRIs
* Patients must be eligible for surgical resection according to the following criteria:

  * Patient competent to sign consent
  * Expectation that the surgeon can resect >= 50% of the Gd-enhancing tumor with low risk of inducing neurological injury
  * Lack of hematologic, cardiac or other medical contraindications to surgery
  * Surgery must take place Monday-Thursday, with the exception of patients being treated at Cleveland Clinic/University Hospitals: these patients may undergo surgery Monday-Friday
  * Patients must have a tumor size ≥ 2.5 cm in diameter in two perpendicular planes in order to enable correlative studies
* Paraffin embedded tissue must be available from initial surgical resection at diagnosis (prior to any treatment)
* Patients may have an unlimited number of prior therapy regimens
* Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

  * 3 months from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not FDA-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., tarceva, hydroxychloroquine, bevacizumab, etc.)
* Patients may be on a non-enzyme-inducing anti-epileptic drug (non-EIAED); they may not be on an EIAED; if previously on an EIAED, patient must be off for at least 14 days prior to the first dose of GDC-0449
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* White blood cells (WBC) ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin ≤ institutional upper limit of normal
* Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤ 4.0 X institutional upper limit of normal
* Creatinine within institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must be able to provide written informed consent
* The effects of GDC-0449 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because Hh signal pathway inhibitors are known to be teratogenic, women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 milli 0international unit/microliter (mL) within 10-14 days prior to treatment start and be required to agree to have the test repeated within 24 hours prior to the first dose of GDC-0449 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of GDC-0449; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of GDC-0449; women of childbearing potential are defined as follows:

  * Patients with regular menses
  * Patients with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
  * Women who have had a tubal ligation
* Women are considered not to be of childbearing potential for the following reasons:

  * The patient has undergone hysterectomy and/or bilateral oophorectomy
  * The patient is post-menopausal defined by amenorrhea for at least 1 year in a woman > 45 years old
* Patients may not be breast-feeding a child
* Patients must have a Mini Mental State Exam score of >= 15

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety, are ineligible
* Patients may not be receiving any other investigational agents
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449 or other agents used in the study are ineligible
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* GDC-0449 inhibits CYP2C8, CYP2C9, and CYP2C19 drug metabolism enzymes in vitro at concentrations that may be clinically relevant; therefore, caution should be exercised when dosing GDC-0449 concurrently with medications that are substrates of CYP2C8, CYP2C9, and CYP2C19 and have narrow therapeutic windows; in addition, GDC-0449 is a substrate of CYP3A4; however, the in vitro metabolic conversion of GDC-0449 is low; effects of CYP inducers (e.g., carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St. John's wort, and troglitazone) on clinical concentrations of GDC-0449 are unknown; likewise, the effects of strong inhibitors of CYP3A4 (e.g., clarithromycin, erythromycin, itraconazole, ketoconazole, nefazodone, and telithromycin) on GDC-0449 clinical concentrations are unknown, and caution should be exercised when dosing GDC-0449 concurrently with inhibitors of CYP3A4
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption are ineligible; patients must be able to swallow capsules
* Patients with clinically important history of liver disease, including viral or other hepatitis or cirrhosis are ineligible
* Patients with a history of uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Patients with uncontrolled intercurrent illness including, but not limited to, hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study because GDC-0449 is an Hh pathway inhibiting agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with GDC-0449, breastfeeding should be discontinued if the mother is treated with GDC-0449
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with GDC-0449

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Nock, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (9):
- United States (9):
  - University of California at Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from March 2010 to April 2011. Subjects were recruited from outpatient cancer centers but all patients needed surgery to participate in this study.
Groups:
- Arm I (Pre-surgery Vismodegib): Patients receive oral Hedgehog antagonist GDC-0449 (vismodegib) once daily for 7 days before therapeutic conventional surgery. Beginning within 28 days after surgical resection, all patients receive oral Hedgehog antagonist GDC-0449 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study; laboratory biomarker analysis
  vismodegib: Given orally
  therapeutic conventional surgery: undergo surgery
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
- Arm II (no Vismodegib Pre-surgery): Patients do not receive treatment before therapeutic conventional surgery. Beginning within 28 days after surgical resection, all patients receive oral Hedgehog antagonist GDC-0449 (vismodegib) once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other: laboratory biomarker analysis
  vismodegib: Given orally
  therapeutic conventional surgery: undergo surgery
  laboratory biomarker analysis: correlative studies
Period: Overall Study
Arm/Group | Arm I (Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery)
Started | 21 | 23
Completed | 20 | 20
Not Completed | 1 | 3
Not completed — no tumor at surgery - treatment effect | 1 | 3

BASELINE CHARACTERISTICS:
Population: 40 patients were evaluable for toxicities, demographics but only 39 for tissue evaluation
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 57 [42 to 79] | 60 [37 to 74] | 59 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 10 | 19
Karnofsky Performance Status Scale [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 80 [60 to 100] | 90 [60 to 100] | 80 [60 to 100]
Mini Mental State Exam (MMSE) [Median (Full Range); unit: units on a scale] — The higher the score the better Range 30 to 0
  units on a scale | 28 [16 to 30] | 29 [16 to 30] | 28 [16 to 30]
Measurable disease [Number; unit: participants]
  Yes | 18 | 18 | 36
  No | 2 | 2 | 4
Number of Prior Treatments [Number; unit: participants]
  1 Prior Treatment | 12 | 15 | 27
  2 Prior Treatments | 6 | 5 | 11
  4 Prior Treatments | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: 6 Months Progression-free Survival (PFS)
Description: Estimated using Kaplan Meier curves. six months calculated from date of treatment onset post-operatively. MRI scan at 6 months must be free of progression Progressive disease Progressive neurological abnormalities not explained by other causes or greater than 25% increase in size of tumor or if new lesion.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I (Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery)
Number analyzed (Participants) | 20 | 20
percentage of patients | 0 [0 to 16.8] | 5 [0.1 to 24.9]

2. Secondary Outcome: Overall Survival Time
Description: The overall failure rate will be estimated along with 95% confidence intervals. A median time of survival will be estimated using standard methods.. Start date based on onset of treatment.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 1(Pre-surgery Vismodegib): Patients receive oral Hedgehog antagonist GDC-0449 (vismodegib) once daily for 7 days before therapeutic conventional surgery.
  Beginning within 28 days after surgical resection, all patients receive oral Hedgehog antagonist GDC-0449 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other: laboratory biomarker analysis
  vismodegib: Given orally
  therapeutic conventional surgery: undergo surgery
  laboratory biomarker analysis: correlative studies
Arm/Group | Arm 1(Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery)
Number analyzed (Participants) | 20 | 20
months | 7.8 [3.7 to 10.2] | 7.6 [5.0 to 13.1]

3. Secondary Outcome: Best Tumor Response Assessed by the Modified Macdonald Radiographic Response Criteria
Description: The Macdonald criteria, roughly similarly to other systems, divides response into 4 types of response based on imaging (MRI) and clinical features
  1: complete response; 2: partial response; 3:stable disease; 4:progression
  Complete response imaging features: disappearance of all enhancing disease (measurable and non-measurable) sustained for at least 4 weeks; no new lesions clinical features; no corticosteroids; clinically stable or improved
  Partial response imaging features: 50% or more decrease of all measurable enhancing lesions sustained for at least 4 weeks: no new lesions clinical features: stable or reduced corticosteroids; clinically stable or improved
  Stable disease imaging features: does not qualify for complete response, partial response or progression clinical features: clinically stable
  Progression imaging features: 25% of more increase in enhancing lesions; any new lesions clinical features: clinical deterioration
Time Frame: evaluated every 8 weeks - 1 year
Population: 3 subjects not evaluable for radiographic response Arm 1 and 4 subjects not evaluable for radiographic response in Arm 2
Measure: Number; unit: participants
Arm/Group | Arm I (Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery)
Number analyzed (Participants) | 20 | 20
participants
  Progressive Disease: number analyzed (Participants) | 17 | 16
  Progressive Disease | 13 | 11
  Stable Disease | 4 | 5

4. Secondary Outcome: Toxicity Incidence Grade 3 or 4 According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
Description: NCI CTCAE grade 3 or 4 possible, probable or definitely related events Grade 3 - severe Grade 4 - life threatening
Time Frame: 30 days from last dose of drug treatment - 1.5 years
Measure: Number; unit: percent of participants
Arm/Group | Arm I (Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery)
Number analyzed (Participants) | 20 | 20
percent of participants
  Lymphocyte count decrase gr3 | 10 | 0
  Stroke gr3 | 5 | 0
  abdominal infection gr3 | 5 | 0
  abdominal pain gr3 | 5 | 0
  atrial flutter gr3 | 5 | 0

5. Secondary Outcome: Incidence of CD133+ Neurospheres by Arm
Description: number of tumor-derived CD133 neurospheres undergoing proliferation and self-renewal
Time Frame: 12 hours post-vismodegib administration
Measure: Number; unit: percent of CD133 Neuospheres
Arm/Group | Arm I (Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery)
Number analyzed (Participants) | 20 | 19
percent of CD133 Neuospheres | 3 | 11

6. Secondary Outcome: Changes in Sonic Hedgehog Pathway Activation
Description: determined by Reverse transcription polymerase chain reaction (RT-PCR) and immunohistochemistry (IHC) (Gli-1, Gli-2, PATCH (PTCH-1b)
Time Frame: Pre-tumor resection and post tumor resection (12 hours)
Population: only small number of samples and thus not enough to give useful information. Samples not processed for outcome and analysis was not performed. No numerical data to report
Arm/Group | Arm 1(Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Determine Drug Effect (Pharmacokinetics) in Plasma for Arm 1
Description: samples collected pre tumor resection (day of surgery) and post-tumor resection (day of surgery
Time Frame: Day of surgery
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | Arm 1(Pre-surgery Vismodegib)
Number analyzed (Participants) | 20
ng/ml
  Plasma | 7638 (1759)
  Intra-tumoral level | 3270 (1326)

ADVERSE EVENTS:
Time Frame: 1year
Description: patients were treated pre and post surgery
Arm/Group | Arm I (Pre-surgery Vismodegib) | Arm II (no Vismodegib Pre-surgery)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pre-surgery Vismodegib) (N=20) | Arm II (no Vismodegib Pre-surgery) (N=20)
abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
anemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 7 (7) | 8 (8)
headache (Nervous system disorders) | 1 (1) | 3 (3)
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lymphocyte count decrease (Investigations) | 2 (2) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — left side
nausea (Gastrointestinal disorders) | 2 (2) | 5 (5)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neutrophile count decrease (Investigations) | 1 (1) | 3 (3)
non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
platelet count decrease (Investigations) | 3 (3) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
stroke (Nervous system disorders) | 1 (1) | 0 (0)
white blood cell decrease (Investigations) | 2 (2) | 4 (4)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less